CLINICAL TRIAL: NCT03981315
Title: Gallbladder Bile Composition in Patients With Gallstones and Healthy Patients
Brief Title: Bile Composition in Healthy and Gallstones Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Son Espases (Other)
Responsible Party: Sponsor
Other Study IDs: BILISGILMOL
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Cholelithiasis; Gall Stone; Gall Bladder Disease
MeSH Terms: conditions — Cholelithiasis; Gallstones; Gallbladder Diseases | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Bile and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lithogenic bile in symptomatic patient: Patients who are performed a cholecystectomy as a treatment of their gallbladder disease
  Interventions: Diagnostic Test: Bile test; Diagnostic Test: Blood test; Diagnostic Test: Gall stone study; Diagnostic Test: Microbiological bile test
- Lithogenic bile in asymptomatic patient: Patients who are performed a cholecystectomy for another reason (cancer, organ donation) and gall stones are found
  Interventions: Diagnostic Test: Bile test; Diagnostic Test: Blood test; Diagnostic Test: Gall stone study; Diagnostic Test: Microbiological bile test
- Non-lithogenic bile: Patients who are performed a cholecystectomy for another reason (cancer, organ donation) without gall stones
  Interventions: Diagnostic Test: Bile test; Diagnostic Test: Blood test; Diagnostic Test: Microbiological bile test

INTERVENTIONS:
Diagnostic Test: Bile test — Analyze bile components related to gall stones synthesis (cholesterol, bile acids, phospholypids, etc.)
Diagnostic Test: Blood test — Analyze blood components related to gall stones synthesis (cholesterol, bile acids, phospholypids, etc.)
Diagnostic Test: Gall stone study — Study of the extracted gall stones, analyzing their composition, type, etc.
  Groups: Lithogenic bile in asymptomatic patient; Lithogenic bile in symptomatic patient
Diagnostic Test: Microbiological bile test — Determination of the microbiological composition of the bile

SUMMARY:
Determine differences between lithogenic and non-lithogenic bile composition.

DETAILED DESCRIPTION:
Gallstones constitute an entity known from antiquity, which have been found even in Egyptian mummies. In elder Greece, Tralliano discovered that gallstones are formed in the liver. Vesalio and Falopio described gallstones inside de gallbladder after a human body dissection and in 1882 Langenbuch performed the first cholecystectomy with good results, becoming the gold standard technique for cholelithiasis.

Nowadays, this pathology represents a public health problem in developed countries due to its high prevalence, which is getting higher, estimated between a 10 and a 15% of the population.

However, gallstones are asymptomatic in the 80% of the cases. In 5 years, a 10-20% of these patients will become symptomatic. The global risk of generating symptoms is about a 2% per year, meanwhile biliary tract complications in asymptomatic patients represent a 0'3% per year.

There are two main types of gallstones. The most common of them (70%) are cholesterol stones, composed of >50% of cholesterol. The other 30% are black pigment stones, with less than 20% of cholesterol in their composition.

The common ways on gallstone formation are: cholesterol supersaturation (due to a liver oversecretion); defects on gallbladder absorption, secretion and motility mechanisms; and higher percentage of deoxycholic acid in the biliary acids due to a slower intestinal movement. All of that leads to supersaturation and cholesterol nucleation.

Black pigment stones are formed of calcium bilirrubinate. The formation mechanism is not clearly defined, but there is an increment in not conjugated bilirubin levels, which is less soluble in water. These gallstones are more frequent in patients who show higher levels of this bilirubin, such as those with hemolysis, Gilbert syndrome or hereditary spherocytosis. They are also common in patients with Crohn disease (specially in those with ileal resection) and cystic fibrosis, in which exists an enterohepatic circulation alteration, driving to an increase on biliary salts and non-conjugated bilirubin levels.

Our work hypothesis is that bile composition in patients with gallstones on the gallbladder is different from those who doesn't show lithiasis.

ELIGIBILITY:
Inclusion Criteria for the Study Group:

1. Patients included for an elective cholecystectomy.
2. Normal hepatic and renal function.
3. Able to understand the nature of the study.
4. Wish to participate in the study and sign the informed consent.

Inclusion Criteria for the Control Group:

1. Patients included for an hepatectomy with gallbladder exeresis for surgery reasons, without lithiasis.
2. Patients included for peritoneal carcinomatosis surgery with gallbladder exeresis for surgery reasons, without lithiasis.
3. Organ donors.
4. Normal hepatic and renal function.
5. Able to understand the nature of the study.
6. Wish to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Under 16 years old
2. Hepatic or renal insufficiency
3. Impossibility to understand the aim of the study

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It includes patients who suffer from gallstones, which are operated for that reason (open or laparoscopic cholecystectomy), and patients who go through the same intervention for other reasons (cancer, organ donation)
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Differences of bile composition between cases and controls | Intra-operatively
  Bilirrubine in mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Son Espases, Palma de Mallorca, Mallorca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibney EJ. Asymptomatic gallstones. Br J Surg. 1990 Apr;77(4):368-72. doi: 10.1002/bjs.1800770405. PMID 2187558
- [Background] Heller F, Bouchier IA. Cholesterol and bile salt studies on the bile of patients with cholesterol gallstones. Gut. 1973 Feb;14(2):83-8. doi: 10.1136/gut.14.2.83. PMID 4696536
- [Background] Jayanthi V, Sarika S, Varghese J, Vaithiswaran V, Sharma M, Reddy MS, Srinivasan V, Reddy GM, Rela M, Kalkura S. Composition of gallbladder bile in healthy individuals and patients with gallstone disease from north and South India. Indian J Gastroenterol. 2016 Sep;35(5):347-353. doi: 10.1007/s12664-016-0685-5. Epub 2016 Sep 16. PMID 27633032
- [Background] Mackay C, Crook JN, Smith DC, McAllister RA. The composition of hepatic and gallbladder bile in patients with gallstones. Gut. 1972 Oct;13(10):759-62. doi: 10.1136/gut.13.10.759. PMID 5087065
- [Background] Reinhold JG, Ferguson LK, Hunsberger A. THE COMPOSITION OF HUMAN GALLBLADDER BILE AND ITS RELATIONSHIP TO CHOLELITHIASIS. J Clin Invest. 1937 May;16(3):367-82. doi: 10.1172/JCI100864. No abstract available. PMID 16694485
- [Background] Shaffer EA. Gallstone disease: Epidemiology of gallbladder stone disease. Best Pract Res Clin Gastroenterol. 2006;20(6):981-96. doi: 10.1016/j.bpg.2006.05.004. PMID 17127183
- [Background] Van Erpecum KJ. Pathogenesis of cholesterol and pigment gallstones: an update. Clin Res Hepatol Gastroenterol. 2011 Apr;35(4):281-7. doi: 10.1016/j.clinre.2011.01.009. Epub 2011 Feb 25. PMID 21353662